CLINICAL TRIAL: NCT04268537
Title: Immunoregulatory Therapy for 2019-nCoV-induced Severe Pneumonia Patients
Brief Title: Immunoregulatory Therapy for 2019-nCoV
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Jianfeng Xie, Director Assistant of ICU, Southeast University, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020YFC0841300-03
Record Dates: First submitted 2020-02-08; First posted 2020-02-13 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: 2019 nCoV, PD-1
Keywords: 2019-ncov; immunotherapy; PD-1; respiratory failure
MeSH Terms: conditions — Parkinson Disease 4, Autosomal Dominant Lewy Body; Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PD-1 group (Experimental): Anti-PD-1 antibody, 200mg, IV, one time
  Interventions: Drug: PD-1 blocking antibody+standard treatment
- thymosin group (Experimental): Thymosin, 1.6 mg sc qd, last for 5 days
  Interventions: Drug: Thymosin+standard treatment
- control group (Placebo Comparator): stand treatment
  Interventions: Other: standard treatment

INTERVENTIONS:
Drug: PD-1 blocking antibody+standard treatment — After randomization, PD-1 blocking antibody 200mg iv, one time. Standard treatment is according to the protocol of treatment of 2019-nCoV infection
  Arms: PD-1 group
Drug: Thymosin+standard treatment — Thymosin 1.6 mg sc qd, last for 5 days. Standard treatment is according to the protocol of treatment of 2019-nCoV infection
  Arms: thymosin group
Other: standard treatment — Standard treatment is according to the protocol of treatment of 2019-nCoV infection
  Arms: control group

SUMMARY:
Sepsis, including viral infections, are major causes of death worldwide. Studies show that in 2017, the number of sepsis patients worldwide reached as high as 48.9 million, of which 11 million patients died. Studies in China also showed that more than 1 million patients died of sepsis in 2015. Previous studies have suggested that sepsis are often secondary to excessive inflammatory response syndrome. However, treatment measures targeting excessive inflammatory response failed to effectively improve the prognosis of patients. PD-1 and PD-L1 are key mediators in T cell depletion in sepsis patients. Therefore, the investigators try to performe a clinical research to investigate the efficacy of PD-1 and thymosin in patients with severe pneumonia associated with lymphocytopenia in 2019 novel coronavirus infection.

DETAILED DESCRIPTION:
Sepsis, including viral infections, are major causes of death worldwide. Studies show that in 2017, the number of sepsis patients worldwide reached as high as 48.9 million, of which eleven million patients died. Studies in China also showed that more than one million patients died of sepsis in 2015. Therefore, how to effectively reduce the mortality of patients with sepsis has become a focus of clinical and basic research.

Previous studies have suggested that sepsis are often secondary to excessive inflammatory response syndrome. However, treatment measures targeting excessive inflammatory response failed to effectively improve the prognosis of patients. The reason is that sepsis-related immune dysfunction can increase the risk of secondary infection and even affect the fatality rate.

The immune checkpoint pathway is the endogenous component of the immune system, which is responsible for checking the immune response and keeping it in a normal physiological state. Tumor cells can evade host recognition through this pathway. One of these immunocheckpoint pathways is the PD-1 and PD-L1 pathways. PD-1 is a receptor expressed on the surface of T cells and ACTS as a negative regulator of T cell function. Monoclonal antibody blocking the activity of PD-1 can successfully reduce tumor load and has been widely used in the clinical treatment of various tumors.

The immune imbalance in patients with sepsis has many similarities tumors. PD-1 and PD-L1 are key mediators in T cell depletion in sepsis patients. Animal models have shown that blocking PD-1 or PD-L1 can prevent T cell death, regulate cytokine production, reduce organ dysfunction and reduce death in sepsis. Previous study showed the clinical safety of anti-PD-1 antibody in sepsis patients through randomized, placebo-controlled trials.

Thymosin has also been proved to regulate cellular immunity in sepsis patients. Some studies have shown that thymosin can significantly reduce the mortality of sepsis patients. At present, phase III clinical research is in progress to further clarify the role of thymosin in patients with sepsis. The purpose of this study was to investigate the efficacy of PD-1 and thymosin in patients with severe pneumonia associated with lymphocytopenia in 2019 novel coronavirus infection.

ELIGIBILITY:
Inclusion Criteria:

1. Adult SARI patients with 2019-ncov infection confirmed by PCR;
2. Absolute value of lymphocytes < 0. 6x 109/L;
3. Severe respiratory failure within 48 hours and requires admission to ICU. (severe respiratory failure was defined as PaO2/FiO2 < 200 mmHg and was supported by positive pressure mechanical ventilation (including non-invasive and invasive mechanical ventilation, PEEP>=5cmH2O))

Exclusion Criteria:

1. Age < 18
2. Pregnant
3. Allergic to experimental drugs
4. The underlying disease is very serious and the expected survival time is less than 6 months (such as advanced malignant tumor);
5. COPD or end-stage lung disease requires home oxygen therapy
6. Expected survival time not exceeding 48 hours
7. Participated in other clinical intervention trials within the last 3 months
8. Autoimmune diseases
9. A history of organ, bone marrow or hematopoietic stem cell transplantation 10. Received radiotherapy and chemotherapy for malignant tumor within 6 months

11.HIV infected patients or diagnosed with acquired immunodeficiency within the past year (CD4 T cells <=200/mm3) 12. Patients receiving anti-hcv treatment 13.90 days of retinal detachment or eye surgery 14. Permanent blindness in one eye 15. History of iritis, endophthalmitis, scleral inflammation or retinitis 16. The competent physician considered it inappropriate to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-02-10 (Estimated); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
lung injury score | 7 days
  proportion of lung injury score decreased 1 or more points

SECONDARY OUTCOMES:
absolute lymphocyte counts | 7, 14 and 28 days
  lymphocyte counts at day 7, 14 and 28 after randimization
serum level of CRP, PCT and IL-6 | 3, 7 and 14 days
  serum level of CRP, PCT and IL-6 at day 3,7 and 14 after randimization
SOFA score | 7 days
  SOFA score at Day 7, with scores range from 0 to 24 and higher score means worse outcome
all cause mortality rate | 28 days
  died at day 28
ventilation free days | 28 days
ICU free days | up to 28 days

IPD SHARING:
Plan to Share IPD: Undecided